CLINICAL TRIAL: NCT03861455
Title: DUPECZEMAIN : Double Blind Placebo-controlled Randomized Multicenter Study Assessing the Efficacy and Safety of Dupilumab in Moderate to Severe Chronic Hands Eczema Refractory to Highly Potent Topical Corticosteroids
Brief Title: Efficacy and Safety of Dupilumab Chronic Hands Eczema Refractory to Highly Potent Topical Corticosteroids
Acronym: DUPECZEMAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/18/0269; 2018-002830-19 (EudraCT Number)
Record Dates: First submitted 2018-11-28; First posted 2019-03-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hand Eczema
Keywords: Chronic Hand Eczema
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive dupilumab 300 mg every 2 weeks after a 600 mg-loading dose of dupilumab on day 0 or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dupilumab group (Experimental): patient receive dupilumab 300 mg every 2 weeks after a 600 mg-loading dose of dupilumab on day 0
  Interventions: Drug: Dupilumab
- placebo group (Placebo Comparator): patient receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dupilumab — patient receive dupilumab 300 mg every 2 weeks after a 600 mg-loading dose of dupilumab on day 0
  Arms: dupilumab group
Drug: placebo — patient receive placebo
  Arms: placebo group

SUMMARY:
Dupilumab has recently demonstrated high efficacy and good safety profile in the treatment of moderate-to-severe atopic dermatitis. There is a crucial need of developing new treatment options in Chronic hand eczema refractory to topical therapy. Investigators hypothesise that Dupilumab will also have high efficacy and good safety profile in the treatment of moderate to severe Chronic hand eczema refractory to highly potent topical corticosteroids.

DETAILED DESCRIPTION:
Chronic hand eczema is a frequent chronic inflammatory skin disease which may have significant physical, psychological and social impact on daily activities, emotional and social life as well as work. In Chronic hand eczema, there is a close relationship between atopic dermatitis (that involves 70% of patients), sensitization to environmental antigens and irritant triggering factors. There are limited treatment options for Chronic hand eczema refractory to highly potent topical steroids. The only systemic treatment labelled in Chronic hand eczema, alitretinoin, is associated with moderate efficacy, high drop-out due to adverse events and it requires strict contraception measures in women of child bearing potential. Dupilumab has recently demonstrated high efficacy and good safety profile in the treatment of moderate-to-severe atopic dermatitis. There is a crucial need of developing new treatment options in Chronic hand eczema refractory to topical therapy. the investigators hypothesise that Dupilumab will also have high efficacy and good safety profile in the treatment of moderate to severe Chronic hand eczema refractory to highly potent topical corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated to a social insurance protection regimen.
* Patients with moderate to severe chronic (>6 months) hand eczema with an Investigator global assessment (IGA) of 3 or 4 (out of a scale of 0 to 4).
* Patients intolerant (according to the physician) or resistant to highly potent topical corticosteroids. Inadequate response (resistance) to highly potent topical corticosteroids is defined as a history of failure to achieve and maintain remission or a low disease activity state (comparable to an IGA score of 0 [indicating clear] to 2 [indicating mild]) despite treatment with a daily regimen of highly potent topical corticosteroids applied for 14 days or for the maximum duration recommended for highly potent topical corticosteroids.
* Patients who are able to understand the study procedures including the ability to complete patient-oriented questionnaires.
* Patients who are able to apply a stable dose of emollients within 7 days before the baseline visit.
* Patients who agree to sign the written informed consent.

Exclusion Criteria:

* Hypersensitivity to dupilumab or to any of its ingredients
* Patients under adult autonomy protection system
* Any other condition (e;g., psoriasis) on the hands that according to the investigator will impair the ability to evaluate treatment effect.
* Treatment with topical corticosteroids or topical calcineurin inhibitors within one week of baseline.
* Treatment with oral immunosuppressants (including cyclosporine, methotrexate, azathioprine, mycophenolate mofetil), alitretinoin or phototherapy within 4 weeks of baseline visit.
* Treatment with an investigational drug within 8 weeks (or 5 half-lives) of baseline.
* Active chronic infection requiring the use of a systemic antibiotic within 2 weeks before study start.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis, aspergillosis) despite infection resolution; or unusually frequent, recurrent, or prolonged infections, per investigator judgment.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Positive for hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody at the screening visit.
* Patients with known helminth infections.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study. Women of childbearing potential who are sexually active and unwilling to use an adequate birth control method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
severity score mTLSS (modified Total Lesion Symptom Score) | Week 16
  The primary outcome measure will be the 16-week percent change since baseline of the severity score mTLSS (modified Total Lesion Symptom Score) The mTLSS combines an evaluation of hand eczema lesions severity including 6 key signs (erythema, desquamation, lichenification/hyperkeratosis, vesiculae, oedema, fissures) and the intensity of pruritus and pain.
  The seven individual CHE symptoms; (erythema, scaling, lichenification or hyperkeratosis, vesiculation, edema, fissures, and pruritus/pain) form the composite scale of mTLSS' strength and each one of them scores from 0 (mild) to 3 (severe). The scores are summed, extending from a base estimation of 0 (no signs or symptoms) to the most extreme of 21 (more serious disease).

SECONDARY OUTCOMES:
Evolution of pruritus | Week 16
  Evolution of pruritus associated with Chronic Hands Eczema at week 16 since baseline measured with a visual analog scale (VAE) from 0 (no itching) to 100 (intense itching).
Evolution of pain | Week 16
  Evolution of pain associated with Chronic Hands Eczema at week 16 since baseline measured with a visual analog scale from 0 (no pain) to 100 (intense skin pain).
Improvement of quality of life | Week 16
  Improvement of quality of life at week 16 since baseline measured by DLQI (Dermatology Life Quality Index) composed of 10 questions (4 possibilities per questions: very much, a lot, a little, not at all).
Improvement of quality of life by EQ-5D-5L | Week 16
  Improvement of quality of life at week 16 since baseline measured by EQ-5D-5L. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his or her current health state using a 0 to 100 mm VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his or her health state by ticking (or placing a cross) in the box associated with the most appropriate statement in each of the 5 dimensions. The VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labeled "best imaginable health state" and "worst imaginable health state." This information can be used as a quantitative measure of health outcome.
evolution of sleep loss | Week 16
  Evolution of sleep loss associated with Chronic Hands Eczema at week 16 since baseline measured with a visual analog scale from 0 (no sleep disorder) to 100 (severe sleep loss).
IGA - Clearance | Week 16
  Clearance or almost clearance of hand eczema at week 16 as defined by an Investigator's global assessment (IGA) of 0 or 1, on a 5 range scale ( from 0 = Clear to 4 = severe disease)
PaGa - Clearance | Week 16
  Clearance or almost clearance of hand eczema at week 16 as assessed by the Patient's global assessment (PaGa) of 0 or 1. The PGA is a single-item question asking the patient how they would rate their overall symptoms. The 5 categories of responses range from "no symptoms"(0) to "severe."(4)
Improvement of work productivity | Week 16
  Improvement of work productivity at week 16 since baseline as assessed by the WPAI questionnaire (Work Productivity and Activity Impairment). The WPAI consists of 6 items grouped into 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. Scores are calculated as impairment percentages, with higher scores indicating greater impairment and less productivity.
Evolution of the Eczema Area and Severity Index (EASI) | Week 16
  Evolution of the Eczema Area and Severity Index at week 16 since baseline in patients who have eczema on other parts of the body than the hands. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Incidence of Treatment-Emergent Adverse Event | Week 16
  The safety throughout the course of the study (at 20 weeks since baseline) by monitoring adverse events, serious adverse events, injection site reactions
evolution of laboratory parameters - full blood count | Week 16
  The evolution of laboratory parameters (full blood count) at week 16 since baseline
evolution of laboratory parameters - transaminases | Week 16
  The evolution of laboratory parameters (transaminase) at week 16 since baseline
evolution of laboratory parameters - total immunoglobulin E | Week 16
  The evolution of laboratory parameters (total immunoglobulin E) at week 16 since baseline
evolution of laboratory parameters - specific immunoglobulin E | Week 16
  The evolution of laboratory parameters (specific immunoglobulin E) at week 16 since baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tauber, Study Director — Lyon Sud Hospital
Locations (4):
- France (4):
  - Saint André Hospital, Bordeaux
  - Hôpital Saint Eloi, Montpellier
  - CHU Lyon-Sud Département d'allergologie et d'immunologie clinique, Pierre-Bénite
  - Larrey Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halioua B. [Hand eczema : disability and impact]. Ann Dermatol Venereol. 2014 Jun;141 Suppl 1:S111-6. doi: 10.1016/S0151-9638(14)70148-6. French. PMID 24953620
- [Background] Cortesi PA, Scalone L, Belisari A, Bonamonte D, Cannavo SP, Cristaudo A, De Pita O, Gallo R, Giannetti A, Gola M, Pigatto PD, Mantovani LG. Cost and quality of life in patients with severe chronic hand eczema refractory to standard therapy with topical potent corticosteroids. Contact Dermatitis. 2014 Mar;70(3):158-68. doi: 10.1111/cod.12130. Epub 2013 Sep 19. PMID 24102212
- [Background] Fowler JF, Graff O, Hamedani AG. A phase 3, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of alitretinoin (BAL4079) in the treatment of severe chronic hand eczema refractory to potent topical corticosteroid therapy. J Drugs Dermatol. 2014 Oct;13(10):1198-204. PMID 25607554
- [Background] Blauvelt A, de Bruin-Weller M, Gooderham M, Cather JC, Weisman J, Pariser D, Simpson EL, Papp KA, Hong HC, Rubel D, Foley P, Prens E, Griffiths CEM, Etoh T, Pinto PH, Pujol RM, Szepietowski JC, Ettler K, Kemeny L, Zhu X, Akinlade B, Hultsch T, Mastey V, Gadkari A, Eckert L, Amin N, Graham NMH, Pirozzi G, Stahl N, Yancopoulos GD, Shumel B. Long-term management of moderate-to-severe atopic dermatitis with dupilumab and concomitant topical corticosteroids (LIBERTY AD CHRONOS): a 1-year, randomised, double-blinded, placebo-controlled, phase 3 trial. Lancet. 2017 Jun 10;389(10086):2287-2303. doi: 10.1016/S0140-6736(17)31191-1. Epub 2017 May 4. PMID 28478972
- [Background] Molin S, Merl J, Dietrich KA, Regauer M, Flaig M, Letule V, Saucke T, Herzinger T, Ruzicka T, Hauck SM. The hand eczema proteome: imbalance of epidermal barrier proteins. Br J Dermatol. 2015 Apr;172(4):994-1001. doi: 10.1111/bjd.13418. Epub 2015 Feb 26. PMID 25244099